CLINICAL TRIAL: NCT06613815
Title: EFFECTIVENESS OF CONVENTIONAL RADIOFREQUENCY OF THE GENICULATED NERVES GUIDED BY SCOPIC VERSUS ULTRASOUND IMAGING FOR THE TREATMENT OF POSTQUIRURGICAL GONALGIA: A RETROSPECTIVE OBSERVATIONAL STUDY
Brief Title: EFFECTIVENESS OF CONVENTIONAL RADIOFREQUENCY OF THE GENICULAR NERVES GUIDED BY SCOPIC VERSUS ULTRASOUND FOR THE TREATMENT OF POSTQUIRURGICAL GONALGIA
Status: Completed | Type: Observational
Sponsor: Fundación Pública Galega Instituto de Investigación Sanitaria. (Other)
Responsible Party: Principal Investigator, ÁLVARO MANUEL GASALLA CADÓRNIGA, Specialist doctor in area, Fundación Pública Galega Instituto de Investigación Sanitaria.
Other Study IDs: nº 2024/211
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritisorconventional Radiofrequencyandgeniculated Nerves
Keywords: knee osteoarthritis, conventional radiofrequency, geniculated nerves, chronic pain.
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- (scopic group, N=19): comparing the analgesic effectiveness of conventional radiofrequency of the geniculate nerves performed in a cohort of patients with a scopy-guided technique (scopic group, N=19)
  Interventions: Other: radiofrequency of the geniculate nerves
- the ultrasound-guided technique (US group, N=38): , comparing the analgesic effectiveness of conventional radiofrequency of the geniculate nerves performed in a cohort of patients with a scopy-guided technique (scopic group, N=19) versus the ultrasound-guided technique
  Interventions: Other: radiofrequency of the geniculate nerves

INTERVENTIONS:
Other: radiofrequency of the geniculate nerves — radiofrequency of the geniculate nerveswith a scopy-guided technique versus the ultrasound-guided technique

SUMMARY:
Knee osteoarthritis is one of the most common joint conditions in the elderly population, characterized by causing pain, stiffness and functional disability in a significant number of cases.

Retrospective, non-randomized observational study, between January 2019 and January 2024, comparing the analgesic effectiveness of conventional radiofrequency of the geniculate nerves performed in a cohort of patients with a scopy-guided technique (scopic group, N=19) versus the ultrasound-guided technique (US group, N=38) in patients referred to the pain unit for chronic gonalgia of moderate-severe intensity after knee surgery.

The main variable studied was the measurement of pain intensity according to the numerical rating scale (NRS) before performing the technique and at 3, 6 and 12 months after radiofrequency denervation of the geniculate nerves.

Conventional radiofrequency of the geniculate nerves of the knee significantly reduces pain intensity over a period of at least 6 to 12 months in patients with chronic postoperative gonalgia, with the ultrasound-guided technique presenting the lowest scores on the numerical pain scale.

It is a simple technique to perform and with few adverse effects, which allows patients to reduce the dose of opioid drugs they take chronically.

DETAILED DESCRIPTION:
Knee osteoarthritis is one of the most common joint conditions in the elderly population, characterized by causing pain, stiffness and functional disability in a significant number of cases.

Retrospective, non-randomized observational study, between January 2019 and January 2024, comparing the analgesic effectiveness of conventional radiofrequency of the geniculate nerves performed in a cohort of patients with a scopy-guided technique (scopic group, N=19) versus the ultrasound-guided technique (US group, N=38) in patients referred to the pain unit for chronic gonalgia of moderate-severe intensity after knee surgery.

The main variable studied was the measurement of pain intensity according to the numerical rating scale (NRS) before performing the technique and at 3, 6 and 12 months after radiofrequency denervation of the geniculate nerves.

The following were measured as secondary variables: the degree of motor block, the reduction in the consumption of opioid drugs, the ease of performing the technique, the degree of patient satisfaction, the appearance of adverse effects and complications related to the technique.

A total of 57 patients were included in the study (19 scopic group and 38 US group). Both techniques were shown to be effective for the control of chronic knee pain. There was a statistically significant reduction in pain intensity at 3, 6 and 12 months (3 [1-5] vs 2 [0-3]; p=0.02 / 3 [2-5] vs 2 [0-3]; p=0.00 / 4 [2-5] vs 2 [1-3]; p=0.00), as well as a reduction in minor opioid requirements (52.6% vs 18.4% p=0.001) in the ultrasound-guided group. No statistical differences were observed between the two groups in terms of the consumption of major opioids or complications of the technique, except for a higher incidence of motor block in the ultrasound-guided group (Bromage scale II: 0% vs 13.2%, p=0.15), which was not clinically relevant.

The degree of patient satisfaction was high in both groups, with no differences being found.Conventional radiofrequency of the geniculate nerves of the knee significantly reduces pain intensity over a period of at least 6 to 12 months in patients with chronic postoperative gonalgia, with the ultrasound-guided technique presenting the lowest scores on the numerical pain scale.

It is a simple technique to perform and with few adverse effects, which allows patients to reduce the dose of opioid drugs they take chronically.

ELIGIBILITY:
Inclusion Criteria:

* people over 18 years of age,physical status ASA I - III, suffering postsurgical chronic Knee pain for more than 3 months, with a baseline pain scale score (NRS) >5 points and failure of other conservative treatments (painkillers, rehabilitation and intraarticular infiltration).

Exclusion Criteria:

* any contraindication for performing regional techniques (infection at the puncture point, alteration of haemostasis, allergy to local anesthetics), pacemaker carriers, non-approval of informed consent, inability to assess postoperative pain, cognitive impairment and known neuropathy of the operated limb.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Due to the reason that it is a retrospective study, sample size calculation was not performed and all patients who underwent this analgesic technique in the last 5 years were consecutively included.
  Continuous quantitative variables were expressed as mean and standard deviation, and the results were contrasted using the Student's T test if data reached normality criteria. Otherwise, they were expressed as median and range and contrasted using the Mann-Whitney U-test. Qualitative variables were expressed in absolute numbers and relative frequencies, and data were contrasted using the Chi square and Fisher's test when necessary. Normality tests were conducted for all continuous quantitative variables. The data were processed using SPSS software version 20.0 (IBM Corporation, Armonk, NY, USA), assuming a p-value below 0.05 as significant.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
The main variable was the measurement of pain intensity assessed by the NRS (Numerical Rating Scale) at different moments: baseline and at 3, 6 and 12 months after performing the technique. | January 2019-January 2024
  The main variable was the measurement of pain intensity assessed by the NRS (Numerical Rating Scale) at different moments: baseline and at 3, 6 and 12 months after performing the technique. As secondary variables, the reduction in opioid requirements were registered.

SECONDARY OUTCOMES:
As secondary variables, the reduction in opioid requirements were registered. | January 2019-January 2024
  As secondary variables, the reduction in opioid requirements were registered.

CONTACTS AND LOCATIONS:
Locations (1):
- Álvaro Manuel Gasalla Cadórniga, Lugo, Spain

IPD SHARING:
Plan to Share IPD: No